CLINICAL TRIAL: NCT01279876
Title: Effects of Melatonin on Clinical and Neuroimaging Indices of Relapsing-Remitting Multiple Sclerosis Patients
Brief Title: Melatonin in Relapsing-Remitting Multiple Sclerosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8153-54-04-87
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Active Comparator)
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator)
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — 3mg oral, daily, one hour before sleep

SUMMARY:
The purpose of this study is to determine whether melatonin is effective in the treatment of relapsing-remitting multiple sclerosis patients as a supplement to the main disease-modifying drugs.

DETAILED DESCRIPTION:
Multiple sclerosis is an autoimmune chronic demyelinating disorder of the central nervous system, and the major cause of disability in the youngsters all over the world, still with no definitely known etiology and treatment. Melatonin is a hormone secreted by pineal gland famous for its role in circadian rhythm regulation, and with known antioxidant effects. It was shown that melatonin is lower in multiple sclerosis patients in the relapse phase in comparison to other diseases and is correlated with the Multiple Sclerosis Functional Composite score of the patients. Melatonin is also suggested to have an immunomodulatory role. Therefore, we hypothesize that melatonin can be effective in the treatment of relapsing-remitting multiple sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* definite diagnosis of relapsing-remitting multiple sclerosis
* EDSS <=5
* at least 6months consumption of interferon beta 1a

Exclusion Criteria:

* illiteracy
* evidence of Nystagmus or visual acuity lower than 5/10 in each of the eyes
* relapse in the last 3 months
* pregnancy or deciding to become pregnant during the following year
* regulatory consumption of warfarin, nifedipine, nonsteroidal anti-inflammatory drugs (NSAIDs), beta-blockers, fluvoxamine, isoniazide, progestin
* history of epilepsy, stroke, major depression, endocrine, hepatic, hematologic, and nephrologic diseases

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-10; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of relapses | one year
EDSS | one year (every 3 months)
  Expanded Disability Status Scale reported by a neurologist
PASAT-3 score | one year (at the beginning and end of the year)
  Paced Auditory Serial Addition Test 3seconds score
proportion of brain gray matter volume to intracranial volume | one year (at the beginning and end of the year)

SECONDARY OUTCOMES:
MSFC score | one year (at the beginning and end of the year)
  Multiple Sclerosis Functional Composite score (Timed 25-foot score + 9-hole peg test score + PASAT-3 score)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hossein Harirchian, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Iranian Center for Neurological Researches, Imam Khomeini Hospital, Tehran, Tehran Province, Iran